CLINICAL TRIAL: NCT03314857
Title: Safety and Effectiveness of Edwards Lifesciences SAPIEN XT Transcatheter Heart Valve in the Chinese Population
Brief Title: China XT: Safety and Effectiveness of Edwards Lifesciences SAPIEN XT THV in the Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015 06
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Aortic Stenosis; Symptomatic Aortic Stenosis; Aortic Regurgitation
Keywords: TAVI; TAVR; CHINA; SAPIEN XT; High Risk; Transcatheter aortic valve implantation; Transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with SAPIEN XT THV (Experimental): Patients will be treated with Edwards SAPIEN XT™ Transcatheter Heart Valve and NovaFlex+ delivery system
  Interventions: Device: SAPIEN XT THV with the NovaFlex+ delivery system

INTERVENTIONS:
Device: SAPIEN XT THV with the NovaFlex+ delivery system — Edwards SAPIEN XT™ Transcatheter Heart Valve along with NovaFlex+ delivery system

SUMMARY:
To evaluate the safety and effectiveness of the SAPIEN XT (Edwards Lifesciences, Irvine, California) transcatheter heart valve implantation (TAVI) in Chinese patients with symptomatic severe calcific aortic stenosis who are considered at high risk for surgical valve replacement.

DETAILED DESCRIPTION:
Edwards SAPIEN XT™ Transcatheter Heart Valve and NovaFlex+ delivery system will be used for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are considered to be operable and high risk for surgical valve replacement: 8 ≤ STS Score ≤ 15 or 15 ≤ Logistic EuroSCORE ≤ 40. If STS score is below 8 and/or Logistic EuroSCORE is below 15, patients should have other clinical or anatomical risk factors that would be considered high risk for surgery and documented by the heart team.
2. Severe symptomatic aortic stenosis requiring aortic valve replacement characterized by one or more of the following within 60 days prior to the index procedure: AVA < 0.8 cm2, Indexed AVA <0.5 cm2/m2, mean gradient > 40mmHg, or peak aortic jet velocity > 4.0m/sec.
3. NYHA Functional Class II or greater.
4. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the EC of the respective clinical site.
5. The study patient agrees to comply with all required post procedure follow-up visits.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment.
2. Aortic valve is a congenital unicuspid or is non-calcified.
3. Aortic valve is bicuspid and the patient is less than 60 years old, or the aortic valve is bicuspid with no raphe (Sievers classification type 0).
4. Anomalous coronary artery that would interfere with proper placement of the valve.
5. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (3):
- China (3):
  - WestChina Hospital, Sichuan University, Sichuan, Chengdu
  - Fuwai Hospital, CAMS&PUMC, Beijing
  - The Second Affiliated Hospital of Zhejiang University School of, Hangzhou

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each study site was allowed up to two roll-in patients. Per the protocol, roll-in patients completed all study visits and procedures but were not part of the analysis. Six of the 67 patients enrolled were roll-in patients.
Groups:
- Patients With SAPIEN XT THV: Patients were implanted with the Edwards SAPIEN XT™ Transcatheter Heart Valve using the NovaFlex+ delivery system.
Period: Overall Study
Arm/Group | Patients With SAPIEN XT THV
Started | 67
Analysis Population (6/67 patients were roll-in patients. Roll-in patients were not included in the analysis.) | 61
Completed | 62 (62/67 patients completed the 30-day primary endpoint visit.)
Not Completed | 5
Not completed — Death | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With SAPIEN XT THV
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (5.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 61
Region of Enrollment [Count of Participants; unit: Participants]
  China | 61
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 6.8 (3.72)
NYHA Class Grouped [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
  Participants
    Class I/II | 5
    Class III/IV | 56

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: All of the deaths that occurred in this population regardless of the cause.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN XT THV
Number analyzed (Participants) | 61
Participants | 4

2. Secondary Outcome: Cardiovascular Mortality
Description: All of the deaths that occurred in this population due to a cardiovascular issue.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN XT THV
Number analyzed (Participants) | 61
Participants | 4

3. Secondary Outcome: Number of Participates With a Stroke
Description: Total number of participates with a stroke.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With SAPIEN XT THV
Number analyzed (Participants) | 61
Participants | 0

ADVERSE EVENTS:
Time Frame: 30-days
Description: All Adverse Events are site-reported.
Arm/Group | Patients With SAPIEN XT THV
All-Cause Mortality (participants affected / at risk) | 4/61
Serious Adverse Events (participants affected / at risk) | 16/61
Other Adverse Events (participants affected / at risk) | 53/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With SAPIEN XT THV (N=61)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial rupture (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2) — These events occurred post procedure and were not associated with device malfunction. "Product issues" is the default MedDRA alignment for device dislocation.
Device failure (Product Issues) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device embolisation (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Vascular access site complication (Injury, poisoning and procedural complications) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Iliac artery perforation (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With SAPIEN XT THV (N=61)
Bundle branch block left (Cardiac disorders) | 11 (11)
Atrioventricular block first degree (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Post procedural fever (Injury, poisoning and procedural complications) | 10 (10)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 9 (9)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 5 (7)
Post procedural constipation (Injury, poisoning and procedural complications) | 4 (4)
Troponin T increased (Investigations) | 28 (28)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6)
Pyrexia (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without the Sponsor's prior written consent, the Principal Investigator shall not publish the clinical study results or any documents containing any Study information at any academic conferences or in any publications of any nature.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03314857/Prot_SAP_000.pdf